CLINICAL TRIAL: NCT00471094
Title: A Phase 2 Study to Evaluate the Safety and Efficacy of Ilaprazole (5 mg QD, 20 mg QD and 40 mg QD) and an Active Comparator, Lansoprazole (30 mg QD) on Healing of Erosive Esophagitis.
Brief Title: Safety and Efficacy of Ilaprazole 5, 20 and 40 mg QD and Lansoprazole 30 mg QD on Healing of Erosive Esophagitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Z-EE05-123; U1111-1127-6202 (Registry Identifier: WHO)
Record Dates: First submitted 2007-05-07; First posted 2007-05-09 (Estimated); Last update posted 2012-02-02 (Estimated); Status verified 2012-01

CONDITIONS: Esophagitis
Keywords: heartburn; erosive esophagitis; healing; population pharmacokinetics; Quality of Life (QoL)
MeSH Terms: conditions — Esophagitis; Heartburn | interventions — ilaprazole; Lansoprazole

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Ilaprazole 5 mg QD (Experimental)
  Interventions: Drug: Ilaprazole
- Ilaprazole 20 mg QD (Experimental)
  Interventions: Drug: Ilaprazole
- Ilaprazole 40 mg QD (Experimental)
  Interventions: Drug: Ilaprazole
- Lansoprazole 30 mg QD (Active Comparator)
  Interventions: Drug: Lansoprazole

INTERVENTIONS:
Drug: Ilaprazole — Ilaprazole 5 mg, capsules, orally, once daily for up to 8 weeks.
  Arms: Ilaprazole 5 mg QD
Drug: Ilaprazole — Ilaprazole 20 mg, capsules, orally, once daily for up to 8 weeks.
  Arms: Ilaprazole 20 mg QD
Drug: Ilaprazole — Ilaprazole 40 mg, capsules, orally, once daily for up to 8 weeks.
  Arms: Ilaprazole 40 mg QD
Drug: Lansoprazole — Lansoprazole 30 mg, capsules, orally, once daily for up to 8 weeks.
  Arms: Lansoprazole 30 mg QD

SUMMARY:
The purpose of this study is to assess the efficacy and safety of 8 weeks of daily treatment with Ilaprazole (5, 20 and 40 mg), once daily (QD), compared to lansoprazole 30 mg in healing subjects with endoscopically proven erosive esophagitis.

DETAILED DESCRIPTION:
This 8 week study will be conducted by approximately 160 investigators in the United States. During this study, esophagitis healing will be evaluated by endoscopy, heartburn and other symptom relief will be evaluated by questionnaire and study drug levels will be measured.

ELIGIBILITY:
Inclusion Criteria:

* Subject must have endoscopically confirmed erosive esophagitis as defined by the Los Angeles (LA) Classification Grading System (A-D).

Exclusion Criteria:

* Evidence of uncontrolled, clinically significant systemic disease; acquired immunodeficiency syndrome (AIDs); a condition likely to require surgery; cancer within 5 years of screening; or abnormal laboratory values.
* Co-existing diseases affecting the esophagus; history of esophageal radiation therapy, cryotherapy, or physiochemical trauma.
* History of esophageal surgery or dilatation of an esophageal stricture other than Schatzki's ring; gastric or duodenal surgery except simple oversew of an ulcer.
* Active gastric or duodenal ulcers or acute upper gastrointestinal hemorrhage within 30 days prior to screening.
* Current or history of Zollinger-Ellison syndrome or other hypersecretory conditions.
* Allergy to any proton pump inhibitor drug (omeprazole, lansoprazole, pantoprazole, rabeprazole, esomeprazole), any component of Ilaprazole, or antacid.
* Unable to tolerate lactose.
* Use of the following medications prior to randomization or anticipated use during the study: proton pump inhibitors, antacids, biphosphonates, histamine (H2) receptor antagonist (examples: Zantac, Tagamet), sucralfate, misoprostol, corticosteroids, prokinetics, Non-steroidal anti-inflammatory drugs (NSAIDs), strong anticholinergics, anticoagulant/anti-platelet aggregate therapy, anticoagulants, digoxin, theophylline, phenytoin.
* History of alcoholism or drug addiction.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 831 (Actual)
Dates: Start 2007-05; Primary Completion 2007-10 (Actual); Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
The crude healing rate of Erosive Esophagitis at week 4 of treatment as assessed by endoscopy. | Week 4

SECONDARY OUTCOMES:
The crude healing rate of Erosive Esophagitis at week 8 of treatment as assessed by endoscopy. | Week 8

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Takeda
Locations (94):
- United States (94):
  - Hueytown, Alabama
  - Huntsville, Alabama
  - Chandler, Arizona
  - Phoenix, Arizona
  - Tempe, Arizona
  - Tucson, Arizona
  - Sherwood, Arkansas
  - Anaheim, California
  - Cypress, California
  - Encinitas, California
  - Garden Grove, California
  - Irvine, California
  - Lancaster, California
  - Mission Hills, California
  - Oakland, California
  - Orange, California
  - Pasadena, California
  - San Diego, California
  - West Covina, California
  - Colorado Springs, Colorado
  - Longmont, Colorado
  - Pueblo, Colorado
  - Bristol, Connecticut
  - Washington D.C., District of Columbia
  - Longwood, Florida
  - Miami, Florida
  - New Smyrna Beach, Florida
  - Pembroke Pines, Florida
  - Tampa, Florida
  - Zephyrhills, Florida
  - Atlanta, Georgia
  - Conyers, Georgia
  - Newnan, Georgia
  - Tucker, Georgia
  - Boise, Idaho
  - Moline, Illinois
  - Rockford, Illinois
  - Clive, Iowa
  - Davenport, Iowa
  - Dubuque, Iowa
  - Wichita, Kansas
  - Metairie, Louisiana
  - Chevy Chase, Maryland
  - Prince Frederick, Maryland
  - Olive Branch, Mississippi
  - Jefferson City, Missouri
  - Kansas City, Missouri
  - Mexico, Missouri
  - Egg Harbor, New Jersey
  - Albuquerque, New Mexico
  - Binghamton, New York
  - Great Neck, New York
  - Rochester, New York
  - Chapel Hill, North Carolina
  - Fayetteville, North Carolina
  - Greensboro, North Carolina
  - Raleigh, North Carolina
  - Wilmington, North Carolina
  - Winston-Salem, North Carolina
  - Cincinnati, Ohio
  - Dayton, Ohio
  - Norman, Oklahoma
  - Oklahoma City, Oklahoma
  - Medford, Oregon
  - Portland, Oregon
  - Beaver Falls, Pennsylvania
  - Harrisburg, Pennsylvania
  - Lansdale, Pennsylvania
  - Warwick, Rhode Island
  - Anderson, South Carolina
  - Charleston, South Carolina
  - Goose Creek, South Carolina
  - Mt. Pleasant, South Carolina
  - Sioux Falls, South Dakota
  - Bristol, Tennessee
  - Chattanooga, Tennessee
  - Johnson City, Tennessee
  - Nashville, Tennessee
  - Amarillo, Texas
  - Austin, Texas
  - Beaumont, Texas
  - Bryan, Texas
  - El Paso, Texas
  - Fort Worth, Texas
  - Houston, Texas
  - Odessa, Texas
  - San Antonio, Texas
  - Midvale, Utah
  - Ogden, Utah
  - Newport News, Virginia
  - Norfolk, Virginia
  - Spokane, Washington
  - Milwaukee, Wisconsin
  - Monroe, Wisconsin